CLINICAL TRIAL: NCT06604650
Title: Community Park-Based Programs for Health Promotion: Active Older Adults Prospective Cohort Study
Acronym: AOA
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Miami-Dade County Parks and Recreation (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00105669_1
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Hypertension; Overweight; Obesity; Cardiovascular Diseases; Sedentary Behavior; Low Physical Fitness
MeSH Terms: conditions — Hypertension; Overweight; Obesity; Cardiovascular Diseases; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Active Older Adults: Body mass index (height and weight), blood pressure and pulse, arm and leg strength and mobility
  Interventions: Behavioral: Active older Adults

INTERVENTIONS:
Behavioral: Active older Adults — The program entails one-hour sessions two or three times per week including aerobic workout, strength training, balance and flexibility exercise delivered online or in-person. Miami-Dade Parks and Recreation is the sponsor of the Active Older Adults prospective cohort study. Duke is conducting a secondary data analysis on data collected as part of the Active Older Adults study.

SUMMARY:
The Active Older Adults prospective cohort study examines the effects of a park-based fitness program on cardiovascular fitness outcomes for older adults (aged 50 years and older). Duke will perform a secondary analysis of the data collected as part of the Active Older Adults prospective cohort study run by Miami-Dade County Parks and Recreation.

DETAILED DESCRIPTION:
The Active Older Adults prospective cohort study examines the effects of a park-based fitness program on cardiovascular fitness outcomes for older adults (aged 50 years and older). Active Older Adults is designed to provide older adults of all fitness levels with physical activity, and aims to promote participant's abilities to maintain independent lifestyles. It is a low-cost, evidence-based group exercise and falls-prevention program. The program entails one-hour sessions two or three times per week including aerobic workout, strength training, balance and flexibility exercise delivered online or in-person. Data are collected at eight Miami Dade Department of Parks, Recreation and Open Spaces (MDPROS) park locations where the program is offered every four months (fall, winter, spring).

Active Older Adults is a park-based fitness program offered by the Miami Dade Department of Parks, Recreation and Open Spaces (MDPROS) that is designed to provide older adults of all fitness levels with physical activity, and aims to promote participant's abilities to maintain independent lifestyles. It is a low-cost, evidence-based group exercise and falls-prevention program. The program entails one-hour sessions two or three times per week including aerobic workout, strength training, balance and flexibility exercise delivered online or in-person. Exercise classes at each park location are offered by bilingual (English/Spanish) licensed instructors and program classes had a consistent format across all parks.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years or older, residing in Miami-Dade County
* All participants enrolled in the Miami-Dade Active Older Adults study will be included in this secondary analysis

Exclusion Criteria:

* Aged less than 50 years, not residing in Miami-Dade County
* Anyone not enrolled in the Miami-Dade Active Older Adults study will be excluded from this secondary analysis

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Active Older Adults is offered in Miami-Dade County (MDC), FL where 40.9% of people older than 65 are sedentary (did not participate in any leisure-time activities, physical activities other than their regular job, during the past month). Within MDC, age-adjusted death rates per 100,000 population (2020-2022) from cardiovascular disease were higher for both Black (291.8.7 vs. 263.4) and Hispanic (179.2 vs. 171.2) residents of MDC vs. statewide, respectively, compared with White (186.2 vs. 198.7) residents. This disparity is particularly relevant for MDC where 69% of people identify as Hispanic or Latino and 17% identify as Black, as opposed to about 19% and 14%, respectively in the United States and 27% and 17% respectively in Florida.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-06-15 (Actual); Primary Completion 2026-06-16 (Estimated); Study Completion 2026-06-16 (Estimated)

PRIMARY OUTCOMES:
Change in Body mass index (height and weight) | Baseline, 12 months, 36 months
Change in blood pressure | Baseline, 12 months, 36 months
Change in arm strength | Baseline, 12 months, 36 months
  Participant arm strength is measured as the total number of arm curls performed in 30 seconds. Participants are seated in a chair while holding a dumbbell or cuff weight (5lb for women and 8lb for men) wrapped around their right or left wrist (the left wrist is employed when the right wrist is impractical).
Change in leg strength | Baseline, 12 months, 36 months
  Leg strength is assessed as the number of chair stands a person could complete in 30 seconds. For one chair stand, participants get up from their seats (with assistance if necessary) and then sit back down.
Change in mobility | Baseline, 12 months, 36 months
  Mobility is measured as the time spent in an Eight-Foot-Up-and-Go test. Participants start seated in a chair, and are instructed to stand up, quickly circle a cone placed eight feet in front of the chair, and then sit back down in the chair. The stopwatch will start when the person fully stands up from the chair and stops when the person sits back down into the chair (recorded in seconds).

CONTACTS AND LOCATIONS:
Overall Officials: Emily D'Agostino, Principal Investigator — Duke University
Locations (1):
- Miami-Dade County Parks, Recreation and Open Spaces Department, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kling HE, D'Agostino EM, Booth J, Hansen E, Hawver E, Mathew MS, Messiah SE. The Feasibility of Collecting Longitudinal Cardiovascular and Fitness Outcomes From a Neighborhood Park-Based Fitness Program in Ethnically Diverse Older Adults: A Proof-of-Concept Study. J Aging Phys Act. 2021 Jun 1;29(3):496-504. doi: 10.1123/japa.2020-0139. Epub 2020 Dec 20. PMID 33348319
- [Background] Kling HE, D'Agostino EM, Booth JV, Patel H, Hansen E, Mathew MS, Messiah SE. The Effect of a Park-Based Physical Activity Program on Cardiovascular, Strength, and Mobility Outcomes Among a Sample of Racially/Ethnically Diverse Adults Aged 55 or Older. Prev Chronic Dis. 2018 Dec 27;15:E166. doi: 10.5888/pcd15.180326. PMID 30589639